CLINICAL TRIAL: NCT02192775
Title: A Phase II Trial of Oncolytic Virotherapy by Systemic Administration of Edmonston Strain of Measles Virus, Genetically Engineered to Express NIS, With Cyclophosphamide, in Patients With Recurrent of Refractory Multiple Myeloma
Brief Title: UARK 2014-21 A Phase II Trial of Oncolytic Virotherapy by Systemic Administration of Edmonston Strain of Measles Virus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 203081
Record Dates: First submitted 2014-07-02; First posted 2014-07-17 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Multiple Myeloma
Keywords: Measles virus; Sodium Iodide Symporter; Cyclophosphamide; Refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MV-NIS + Cyclophosphamide (Experimental)
  Interventions: Drug: MV-NIS

INTERVENTIONS:
Drug: MV-NIS — one dose in conjunction with a 4 day course intravenously
  Other Names: Recombinant Edmonston measles virus with human NIS gene

SUMMARY:
The purpose of this study is to determine the clinical efficacy of MV-NIS (measles virus-sodium iodide symporter) therapy for people with relapsed/refractory myeloma when given with cyclophosphamide

DETAILED DESCRIPTION:
The drug used in this trial is a modified version of the measles virus used to vaccinate children. The virus has been altered by having an extra gene (piece of DNA) added to it to allow a protein called NIS to be inserted into it. NIS is normally found in the thyroid gland ( a small gland in the neck) and helps the body concentrate iodine. Having this additional gene will make it possible to track where the virus goes in the body.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed patients must have a confirmed MM diagnosis with high-risk disease as defined by GEP70 risk score ≥ 0.66 or GEP80 gene score of ≥ 2.48 or metaphase cytogenetic abnormalities or LDH ≥ 360 U/L due to MM (Rule out hemolysis, infection and contact PI for clarification if any doubt). Patients must have relapsed after auto-PBSCT followed by further chemotherapy
* ≥2 months must have elapsed after the last peripheral blood stem cell transplant prior to enrollment
* Zubrod ≤ 2, unless solely due to symptoms of MM-related (bone) disease
* Patients must have a platelet count of ≥ 20,000/µL within 45 days of registration, unless lower levels are explained by extensive BM plasmacytosis or extensive prior therapy
* Patients must be at least 18 years of age and not older than 75 years of age at the time of registration
* Participants must have preserved renal function as defined by a serum creatinine level of ≤ 3 mg/dL within 45 days of registration
* Participants must have an ejection fraction by ECHO or MUGA scan ≥ 40% within 45 days prior to registration
* Patients must have adequate pulmonary function studies > 50% of predicted on mechanical aspects (FEV1, etc) and diffusion capacity (DLCO) > 50% of predicted within 45 days prior to registration. If the patient is unable to complete pulmonary function tests due to MM related pain or condition, exception may be granted
* Patients must have signed an IRB-approved informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization form
* Patients must have anti-MV IgG titer of ≤ 0.5U/mL (Mayo clinic assay). Mayo Clinic will also assay the patients' IgM titer and perform a neutralizing antibody plaque-assay to determine recent MV exposure and the ability of the patients' circulating antibodies to inhibit MV propagation on Vero cells, respectively. While these tests are additional indicators of patient eligibility, final enrollment decision will be determined by IgG levels

Exclusion Criteria:

* Patients may not be positive for the Human Immunodeficiency Virus (HIV)
* History of poorly controlled hypertension, diabetes mellitus, or any other serious medical illness or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol or could be considered to be an exclusion criterion deemed by the PI
* Patients must not have prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has not received treatment for one year prior to enrollment. Other cancers will only be acceptable if the patient's life expectancy exceeds three years as determined by the PI
* Pregnant or nursing women may not participate. Women of childbearing potential must have a negative pregnancy test documented within one week of registration. Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* Exposure to household contacts ≤ 15 months old or household contact with known immunodeficiency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frits Van Rhee, MD, Ph.D, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Science, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MV-NIS + Cyclophosphamide
Started | 2
Completed | 0
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | MV-NIS + Cyclophosphamide
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: The Effectiveness of MV-NIS Therapy as Measured by the International Myeloma Working Group (IMWG) Guidelines
Description: The primary objective of this study is to assess the effectiveness of MV-NIS therapy for people with relapsed/refractory myeloma when given with cyclophosphamide
Time Frame: 1 year
Population: Only two subjects were enrolled. Both passed away while enrolled. No data were collected.
Arm/Group | MV-NIS + Cyclophosphamide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | MV-NIS + Cyclophosphamide
All-Cause Mortality (participants affected / at risk) | 2/2
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MV-NIS + Cyclophosphamide (N=2)
Hyperammonia (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Decreased Respiratory Rate (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acidosis (Metabolic) (Metabolism and nutrition disorders) | 1 (1)
Alterned Mental State (Nervous system disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MV-NIS + Cyclophosphamide (N=2)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Localized Edema (General disorders) | 1 (1)
Neutrophil Count Decreased (Investigations) | 2 (3)
C-Reactive Protein Increased (Investigations) | 2 (2)
Lactate Increased (Investigations) | 1 (1)
Lactate Dehydrogenase Increased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Enterocolitis Infectious (Infections and infestations) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 1 (2)
White Blood Count Decreased (Investigations) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-21): https://cdn.clinicaltrials.gov/large-docs/75/NCT02192775/Prot_SAP_000.pdf